CLINICAL TRIAL: NCT04503122
Title: Baroreflex Sensitivity in Patients Undergoing Atrial Fibrillation Ablation: Association With Arrhythmia Recurrences
Brief Title: Baroreflex Sensitivity in Patients Undergoing Ablation of Atrial Fibrillation
Acronym: BARO-AF
Status: Completed | Type: Observational
Sponsor: Poitiers University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: BARO-AF
Record Dates: First submitted 2020-08-03; First posted 2020-08-07 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-12

CONDITIONS: Paroxysmal Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: pulmonary vein isolation — pulmonary vein isolation : cryoablation or radiofrequency

SUMMARY:
Atrial fibrillation is the most common arrhythmia. The posterior surface of the left atrium is covered by an extensive network belonging to the autonomic nervous system that can be damaged during the ablation. The involvement of the autonomous nervous system in the genesis and maintenance of atrial fibrillation remains poorly understood. Baroreflex sensitivity is a non-invasive method assessing autonomous nervous system activity.

The rate of atrial fibrillation recurrence after ablation is currently high and a better understanding of the mechanisms associated with recurrence is essential to improve selection of the patients who will benefit the most from this procedure.

The aim of this study is to evaluate the association between the baroreflex sensitivity and atrial fibrillation recurrences and to analyze the prognostic contribution of the baroreflex measurement compared to other published criteria.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years old,
* Patients with paroxysmal atrial fibrillation, hospitalized for atrial fibrillation ablation,
* Assessable baroreflex sensitivity before ablation,
* Free subject, without guardianship or curatorship or subordination,
* Patients benefiting from a Social Security assurance,
* Informed consent signed by the patient after clear and fair information about the study.

Exclusion Criteria:

* Age < 18,
* History of atrial fibrillation ablation,
* Inability to calculate the baroreflex sensitivity
* Contraindication to the performance of a cardiac CT scan (allergy to iodine, severe renal insufficiency with clearance <30 ml/mn/m2),
* Inability to have continuous ECG recording by subcutaneous Holter,

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients with paroxysmal atrial fibrillation undergoing atrial fibrillation ablation
Sampling Method: Probability Sample
Enrollment: 116 (Actual)
Dates: Start 2021-06-22 (Actual); Primary Completion 2025-11-13 (Actual); Study Completion 2025-11-13 (Actual)

PRIMARY OUTCOMES:
Mean slope assessed before ablation in the recurrence and the non-recurrence groups | Recurrence is assessed at one year of follow-up
  To compare baroreflex sensitivity assessed by mean Slope 1 month before the ablation in the recurrence group at 1 year and in the no AF recurrence group at 1 year.

SECONDARY OUTCOMES:
Association between baroreflex sensitivity assessed before ablation and atrial fibrillation burden | Burden is assessed at one year of follow-up
  Association between baroreflex sensitivity evaluated by mean slope, LF gain and HF gain 1 month before AF ablation and AF burden after 1 year of follow-up;
Baroreflex sensitivity fall between the groups with and without AF recurrence | Recurrence is assessed at one year of follow-up
  To compare the baroreflex sensitivity fall between before and day1 of ablation between the groups with and without AF recurrence at 1 year follow-up ;
Evolution of baroreflex sensitivity | Before, day 1 and month 3 after the ablation
  To describe the evolution of baroreflex sensitivity in the group with and in the group without recurrence.
Biological and imaging parameters | Burden is assessed at one year of follow-up
  To look for an association between biological and imaging parameters and atrial fibrillation burden at 1 year.
Quality of life | before and at one year after atrial fibrillation ablation
  To compare quality of life before and at one year after atrial fibrillation ablation in patients with and without AF recurrence;

CONTACTS AND LOCATIONS:
Locations (1):
- CHU de Poitiers, Poitiers, France

IPD SHARING:
Plan to Share IPD: Undecided